CLINICAL TRIAL: NCT04811014
Title: Houston Emergency Engagement System for Youths and Adolescents
Brief Title: Young Houston Emergency Opioid Engagement System
Acronym: YHEROES
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, James Langabeer, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-20-1376
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Opioid-use Disorder; Opioid Dependence; Opioid Overdose; Opioid Use; Substance Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Therapeutics; Self-Help Groups; Psychotherapy, Group; Community-Institutional Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MOUD induction and behavioral interventions among opioid-dependent youths (Experimental): Induction into medication for opioid use disorder (MOUD) treatment and behavioral interventions
  Interventions: Drug: Buprenorphine, Naloxone Drug Combination; Behavioral: Individual Counseling; Behavioral: Peer Recovery Support Services; Behavioral: Support Group; Behavioral: Referral to Medication Management; Behavioral: Assertive Outreach

INTERVENTIONS:
Drug: Buprenorphine, Naloxone Drug Combination — 8mg of buprenorphine/2mg of naloxone to initiate MOUD treatment and bridge, if necessary, until referral to MOUD clinic can be made for ongoing treatment
  Other Names: Suboxone
Behavioral: Individual Counseling — One-on-one counseling with a licensed chemical dependency counselor
  Other Names: Therapy
Behavioral: Peer Recovery Support Services — 24/7 support from our team of certified peer recovery support specialists to assist with emotional support and case management
  Other Names: Peer Coaching; Recovery Coaching
Behavioral: Support Group — Referrals to youth-focused support groups and eventual creation of in-house youth-focused support groups
  Other Names: Group Therapy
Behavioral: Referral to Medication Management — Study staff will refer patients to long-term MOUD providers in the community
Behavioral: Assertive Outreach — The investigators will conduct weekly outreach to youths who experienced an opioid overdose and attempt to initiate treatment. Outreach is completed by a paramedic and peer coach.
  Other Names: Community Outreach

SUMMARY:
The Houston Emergency Response Opioid Engagement System for Youths and Adolescents (Young HEROES) is a community-based research program integrating assertive outreach, medication for opioid use disorder (MOUD), behavioral counseling, and peer recovery support. The objective is to compare differences in engagement and retention in treatment for individuals with opioid use disorder. The investigators also intend to understand the prevalence of opioid overdoses and OUD among youth in Houston.

DETAILED DESCRIPTION:
The Houston Emergency Response Opioid Engagement System for Youths and Adolescents (Young HEROES) is a non-randomized cohort study based at the University of Texas Health Science Center of Houston. This study recruits participants through three avenues: assertive community outreach with a peer coach and paramedic following and opioid overdose, community referrals, and emergency department referrals. The study explores the effect of the combination of assertive outreach, same-day induction into medication for opioid use disorder, ongoing maintenance treatment, behavioral counseling, peer recovery support, and paramedic follow-up on patient outcomes. The primary outcome is engagement and retention in outpatient treatment. Secondary outcomes include quality of life assessment as well as subsequent relapses and overdoses. The hypothesis is that patients with earlier induction into MOUD treatment who receive routine follow-up, are more likely to engage and remain in treatment long-term.

ELIGIBILITY:
Inclusion Criteria:

* In otherwise good health based on physician assessment and medical history
* Drug screen positive for opioids
* Patients express a willingness to stop opioid use
* Meet Diagnostic and Statistical Manual of Mental Disorders - Text Revision (DSM-IV-TR) criteria for opioid dependence
* Patients must be able to speak English
* Be agreeable to and capable of signing the informed consent and assent (parent or guardian must consent, minor must assent)

Exclusion Criteria:

* Non-English-speaking patients
* Have a known sensitivity to buprenorphine or naloxone
* Be physiologically dependent on alcohol, benzodiazepines, or other drugs of abuse that require immediate medical attention. Other substance use diagnoses are not exclusionary.
* Have a medical condition that would, in the opinion of the study physician, make participation medically hazardous, including unstable cardiovascular disease, neurological deficits, trauma, acute hepatitis, stroke, and liver or renal disease)
* Be acutely psychotic, severely depressed, and in need of inpatient treatment, or is an immediate suicide risk
* Be a nursing or pregnant female

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient retention in treatment | 30 days after enrollment
  Percentage of enrolled youth in treatment over time
Patient abstinence from opioids | 30 days after enrollment
  Days without substance use

SECONDARY OUTCOMES:
Frequency of opioid emergencies among adolescents in Houston, Texas | Through study completion, an average of 3 years
  Prevalence of opioid overdoses among youth

CONTACTS AND LOCATIONS:
Overall Officials: James R Langabeer, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States